CLINICAL TRIAL: NCT03691389
Title: Investigating the Relationship Between Children With ADHD and Conduct Disorder and Their Parents in Reduction of Symptoms
Brief Title: Investigating the Relationship Between Parents and Their Children With ADHD and Conduct Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: YNC-SASSI-Quali
Record Dates: First submitted 2018-09-22; First posted 2018-10-01 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Observation

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to uncover mechanisms of action underlying any long-term change in youth antisocial behavior by considering the role of child and family characteristics as mediators and moderators of change. The study design is qualitative interviews to be conducted face-to-face with parents of children previously diagnosed with Conduct Disorder and Attention Deficit Hyperactivity Disorder (ADHD) but no longer meet diagnostic criteria. Questions will be asked to understand participants' parenting experience over time (before, during and after their children's treatment).

ELIGIBILITY:
Inclusion Criteria:

* Parents of children who participated in previous study "Supplements and Social Skills Intervention" conducted by Singapore Institute of Mental Health Child Guidance Clinic.
* Children no longer meet the criteria for Conduct Disorder and ADHD, as measured by Antisocial Process Screening Device (APSD) Callous-Unemotional score of 7 or less, and who do not meet the cut-off for rule-breaking and aggressive behavior determined by Child Behavior Checklist (CBCL). These data were collected from a previous study.

Exclusion Criteria:

* Children who still meet the requirements of Conduct Disorder and ADHD as defined above.
* Parents who did not indicate that they wish to be contacted for follow-up studies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists parents of children who participated in a previous longitudinal study that investigates the effectiveness of omega-3 supplementation and social skills training in treating Conduct Disorder and Attention Deficit Hyperactivity Disorder (ADHD). The study ended noting that some children no longer meet the criteria of the disorders and based on existing literature, parental interactions may have a role in this phenomenon. As such, this research proposes to interview parents of these children to understand more.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Parental style and interactions with children | 1 year
  Qualitative interview based on a phenomenological analysis will seek to understand from parents before, during, and after the treatment (previous intervention) about their interactions with their children, especially when problematic behavioural issues occur. All interviews were transcribed verbatim as much as possible, then subjected to a first round of open coding through identification of words, sentences or paragraphs expressing common ideas. Thereafter, a framework of themes was derived and interview content was organized systematically for analysis. The transcripts will also be rotated among researchers for the various stages of coding, such that each transcript was coded by at least two different people. This was to minimize subjectivity in coding and ensure the inter-rater consistency of the codes.